CLINICAL TRIAL: NCT03997812
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VVZ-149 Injections for the Treatment of Postoperative Pain Following Bunionectomy
Brief Title: Evaluate the Efficacy and Safety of VVZ-149 Injections for the Treatment of Postoperative Pain Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVZ149-POP-P2-US004
Record Dates: First submitted 2019-05-28; First posted 2019-06-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VVZ-149 Injections (Experimental)
  Interventions: Drug: VVZ-149 Injections
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149 Injections — IV infusion of 1000 mg of VVZ-149
  Other Names: Opiranserin Injections
  Arms: VVZ-149 Injections
Drug: Placebo — IV infusion of 0 mg of VVZ-149
  Arms: Placebo

SUMMARY:
The purpose of this phase 2 study is to evaluate the efficacy and safety of an analgesic drug candidate, VVZ-149 Injections for treating post-operative pain following bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women must be between the ages of 18 to 70 years, inclusive. Female subjects must meet additional criteria in relation to childbearing potential.
* Subjects must be undergoing a planned bunionectomy without collateral procedures.
* Subjects must have the ability to provide written informed consent.
* Subjects must have the ability to understand study procedures and communicate clearly with the Investigator and staff.
* Subjects must be classified as American Society of Anesthesiologists risk class I to II.

Exclusion Criteria:

* Subjects undergoing emergency or unplanned surgery.
* Subjects undergoing a repeat operation.
* Subjects with pre-existing conditions (other than bunion) causing preoperative pain at the site of surgery.
* Female subjects who are pregnant or breastfeeding.
* Diagnosis of chronic pain and ongoing or frequent use of pain medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Total Area Under the Curve (AUC) of Pain Intensity for 12 hours after the start of study drug infusion | 0-12 hours after the start of study drug infusion
  Using Numeric Pain Rating Scale (NRS, 0-10 at rest)

SECONDARY OUTCOMES:
AUC of pain intensity for 24 hours after the start of study drug infusion. | 0-24 hours after the start of study drug infusion
Total opioid consumption up to 12 hours after the start of study drug infusion. | 0-12 hours after the start of study drug infusion
Total opioid consumption up to 24 hours after the start of study drug infusion. | 0-24 hours after the start of study drug infusion
Percentage of cumulative subjects that used rescue medication prior to each scheduled pain intensity assessment time point. | 0-24 hours after the start of study drug infusion
Time until the subject requested first and second rescue medications. | 0-24 hours after the start of study drug infusion
Time to perceptible, meaningful, and confirmed perceptible pain relief. | 0-12 hours after the start of study drug infusion

CONTACTS AND LOCATIONS:
Overall Officials: Doo Lee, PhD, Study Chair — Vivozon, Inc.
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, Anaheim, California
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No